CLINICAL TRIAL: NCT02010723
Title: Comparison of Surgery Versus Foam Sclerotherapy for Isolated Accessory Great Saphenous Vein Varicosis
Brief Title: Surgery Versus Sclerotherapy for Isolated Accessory Great Saphenous Vein Varicosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kornelia Boehler, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060508; 255/2006 (Other: Ethikkommission medical university of vienna)
Record Dates: First submitted 2013-11-18; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Varicose Veins
Keywords: varicosis; foam sclerotherapy; surgery
MeSH Terms: conditions — Varicose Veins | interventions — Surgical Procedures, Operative; Sclerotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery (Active Comparator): crossectomy and avulsion of the varicose anterior accessory great saphenous vein (AAGSV) under local anesthesia
  Interventions: Procedure: surgery
- sclerotherapy (Experimental): foam sclerotherapy with aethoxysclerol foam
  Interventions: Drug: sclerotherapy with aethoxysclerol foam

INTERVENTIONS:
Procedure: surgery — crossectomy and avulsion of the varicose anterior accessory great saphenous vein (AAGSV) under local anesthesia
  Arms: surgery
Drug: sclerotherapy with aethoxysclerol foam — foam sclerotherapy with aethoxysclerol foam
  Arms: sclerotherapy

SUMMARY:
The purpose of this study is to compare two therapeutic procedures in the treatment of isolated varicosis of the anterior accessory great saphenous vein (AAGSV): crossectomy and avulsion of the varicose AAGSV versus foam sclerotherapy of the AAGSV.

ELIGIBILITY:
Inclusion Criteria:

* reflux in anterior accessory great saphenous vein (AAGSV) > 0,5 sek

Exclusion Criteria:

* concomitant reflux in great saphenous vein (GSV)
* reflux in the deep venous system (postthrombotic syndrome)
* acute thrombosis
* hypercoagulability
* allergy to aethoxysclerol or local anesthetics
* immobility
* open foramen ovale
* bacterial infection of the skin
* pregnancy and breast feeding
* peripheral arterial occlusive disease III, IV (PAOD)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
duplex-sonographic recurrence after 3 years | 3 years
  duplex-sonographic recurrence is defined as reverse blood flow of > 0.5 sec along the anterior accessory great saphenous vein (AAGSV) in the sclerotherapy group or in new anterior thigh varicosities connected to the previous saphenofemoral junction (NATV) in the surgical group.

SECONDARY OUTCOMES:
duplex-sonographic recurrence after 1 year | 1 year
  duplex-sonographic recurrence is defined as reverse blood flow of > 0.5 sec along the AAGSV in the sclerotherapy group or in new anterior thigh varicosities connected to the previous saphenofemoral junction (NATV) in the surgical group
clinical recurrence | 1 year and 3 years
  Clinical recurrence is evaluated by determination of the current Clinical-Etiology- Anatomy- Pathophysiology (CEAP) classification and reappearance of new varicose veins in the treated area
neovascularisation in the saphenofemoral junction | 1 year and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kornelia Boehler, MD, Principal Investigator — Medical University of Vienna, University Clinic of Dermatology, Department of General Dermatology
Locations (1):
- Medical University of Vienna, Department of General Dermatology, Vienna, Vienna, Austria

REFERENCES:
- [Background] Prinz N, Selzle K, Kamionek I, Sagoo KS, Leberig A, Kaiser R, Schonath M. [Surgery of the lateral accessory saphenous vein]. Zentralbl Chir. 2001 Jul;126(7):526-7. doi: 10.1055/s-2001-16280. German. PMID 11503465
- [Background] Breu FX, Guggenbichler S, Wollmann JC; Second European Consensus Meeting on Foam Sclerotherapy. Duplex ultrasound and efficacy criteria in foam sclerotherapy from the 2nd European Consensus Meeting on Foam Sclerotherapy 2006, Tegernsee, Germany. Vasa. 2008 Feb;37(1):90-5. doi: 10.1024/0301-1526.37.1.90. PMID 18512547
- [Background] Theivacumar NS, Darwood RJ, Gough MJ. Endovenous laser ablation (EVLA) of the anterior accessory great saphenous vein (AAGSV): abolition of sapheno-femoral reflux with preservation of the great saphenous vein. Eur J Vasc Endovasc Surg. 2009 Apr;37(4):477-81. doi: 10.1016/j.ejvs.2008.11.035. Epub 2009 Feb 7. PMID 19201621